CLINICAL TRIAL: NCT07203898
Title: A Phase 1, Open-Label, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of IPM514 in Patients With Unresectable Advanced, Recurrent or Metastatic Esophageal Squamous Cell Carcinoma (ESCC).
Brief Title: A Study of IPM514 in Patients With Esophageal Squamous Cell Carcinoma.
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Immupeutics Medicine Technology Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPM514-002
Record Dates: First submitted 2025-09-22; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IPM514 (Experimental)
  Interventions: Biological: IPM514

INTERVENTIONS:
Biological: IPM514 — 2 primary immunization cycles: IPM514 will be administered once a week (QW) for 3 consecutive doses per cycle, there will be a 2-week interval between the two cycles.
  Maintenance treatment: 6 doses administered every 3 weeks (Q3W), and 4 doses administered every 6 weeks (Q6W), if treatment continuously benefit the participant.

SUMMARY:
This is a Phase 1, open-label, multicenter study to assess the safety, tolerability, and preliminary efficacy of IPM514 in patients with unresectable advanced, recurrent or metastatic esophageal squamous cell carcinoma.

IPM514 will be administered by intramuscular injection. Six ascending dose cohorts of IPM514 will be evaluated, with each cohort planned to enroll 3-6 qualified participants after a screening period of up to 28 days, following 3 + 3 study design format, the dose levels are as follows: 50 µg, 100 µg, 200 µg, 300 µg, 450 µg, and 600 µg. It may be adjusted during the dose escalation study based on the emerging data of safety, efficacy, and biological responses upon Safety Monitoring Committee (SMC) approval.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate in this study, a patient must meet all the following criteria:

  1. Male or female, aged ≥ 18 years on the day the patient voluntarily agrees to participate in the study.
  2. Able to provide written informed consent and can understand and agree to comply with the requirements of the study and the schedule of assessments.
  3. Histologically confirmed diagnosis of ESCC.
  4. Patients' prior systemic therapy must have included at least a PD-1/PD-L1 inhibitor and a platinum-based chemotherapy regimen and have disease progression confirmed by imaging during or after these treatments.

     NOTE:

     • Patients with disease progression that occurs during treatment or within 6 months of cessation of neoadjuvant/adjuvant treatment, this neoadjuvant/adjuvant treatment will be regarded as a line of systemic treatment.
  5. At least one measurable/evaluable lesion by RECIST v1.1 as determined by local site investigator/radiology assessment within 28 days prior to first dose.

     NOTE: Lesions that have been previously irradiated may be considered evaluable provided there is evidence of disease progression following the completion of radiation therapy.
  6. The HLA typing is HLA-A*02:01 and/or HLA-A*11:01.
  7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
  8. Life expectancy ≥12 weeks.
  9. The organ function level in the screening period must meet the following requirements (Laboratory data will not be valid if the patient has received growth factors or blood transfusion for prophylactic use within 7 days before the laboratory testing):

     * Absolute neutrophil count (ANC) ≥ 1500 cells/mm3
     * Platelet count （PLT）≥ 100,000 cells/mm3
     * Hemoglobin（Hb）≥ 90 g/L
     * Serum creatinine (Cr) ≤ 1.5 × upper limit of normal (ULN) and Creatinine clearance rate (Cockcroft-Gault Formula) ≥ 50 mL/min
     * Serum total bilirubin ≤1.5 × ULN (or < 3 × ULN in patients with Gilbert's syndrome or patients with liver metastasis)
     * Aspartate transaminase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN (or ≤ 5.0 × ULN in patients with liver metastases)
     * Prothrombin time (PT), International normalized ratio (INR) ≤ 1.5 × ULN unless the patient is receiving anti-coagulant therapy
     * Urine routine/24-hour urine protein quantification: Urine protein qualitative ≤ 1+ (if urine protein qualitative ≥ 2+, then 24-hour urine protein < 1 g can be enrolled)
     * Serum albumin ≥ 28 g/L.
  10. Prior chemotherapy, radiotherapy, immunotherapy or any investigational therapies used to control cancer, all AEs have either returned to baseline or Grade 0~1, and stabilized.
  11. Females of childbearing potential (WOCBP) must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) at screening. Patients that are postmenopausal (with spontaneous amenorrhea for at least 24 months) or permanently sterilized can be considered as not having reproductive potential. Female patients of reproductive potential must agree to use highly effective contraception during and for 3 months after the last trial drug administration.
  12. Non-sterile males who have female sexual partner(s) of childbearing potential must use highly effective form of birth control for the duration of the study, and for at least 3 months after the last trial drug administration.

      * A sterile male is defined as one for whom known azoospermia, in a semen sample examination, has been previously demonstrated as definitive evidence of infertility.
      * Males with known 'low sperm counts' (consistent with 'sub-fertility') are not to be considered sterile for purposes of this study.

Exclusion Criteria:

* To be eligible to participate in this study, a patient cannot meet any of the following exclusion criteria:

  1. Known allergy to the components of the study drug.
  2. Esophageal squamous cell carcinoma known to be prone to complete obstruction under endoscopy requires interventional therapy to relieve the obstruction.
  3. After stent implantation in esophagus or trachea, patients who are at high risk of bleeding or perforation due to significant tumor invasion of adjacent organs (aorta or trachea), or who have developed fistulas.
  4. Uncontrollable pleural effusion, pericardial effusion, or ascites requiring frequent drainage (recurrence within 2 weeks of intervention).
  5. Active leptomeningeal disease or uncontrolled brain metastasis. Patients with a history of treated and, at the time of screening, stable central nervous system (CNS) metastases are eligible, provided they meet all the following:

     * Brain imaging at screening shows no evidence of interim progression, clinically stable for at least 4 weeks and have no evidence of new brain metastases.
     * Have measurable and/or evaluable disease outside the CNS.
     * No ongoing requirement for corticosteroids as therapy for CNS disease; off steroids 14 days prior to first dose.
     * No stereotactic radiation or whole-brain radiation within 14 days prior to the first dose.
  6. With previous history of other malignant tumors, except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix or breast.
  7. With a local infection or systemic infection which requires systemic antibiotic treatment within 2 weeks prior to the first dose of trial treatment.
  8. With a history of splenectomy, or congenital asplenia.
  9. Patients who have had major surgery (e.g., requiring general anesthesia) within 4 weeks before screening, have not fully recovered from surgery, or have a surgery planned during the time of trial participation.
  10. Has active autoimmune disease or history of autoimmune diseases at high risk of relapse.

      NOTE: Patients with following diseases may be enrolled if they meet all other eligibility criteria: controlled type I diabetes, hypothyroidism managed with hormone replacement therapy only, controlled celiac disease, skin diseases not requiring systemic treatment (such as vitiligo, psoriasis, or alopecia), or diseases not expected to recur in the absence of external triggering factors.
  11. Has a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days prior to first dose:

      * Patients who have a history of organ transplant, including stem cell allograft are not permitted to enroll.
      * Adrenal replacement steroid dose ≤ 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
      * Patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption).
      * A brief course of corticosteroids for prophylaxis (eg, contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
  12. Has received:

      * Within 28 days or 5 half-lives (whichever is shorter but at least 14 days) of the first study drug administration: any anti-tumor drug therapy, such as chemotherapy, targeted therapy, immunotherapy, and biological therapy, or any investigational therapy.
      * Within 14 days of the first study drug administration: any Chinese herbal medicine or Chinese patent medicines used to control cancer or boost immunity.
      * Within 14 days of the first study drug administration: palliative radiation treatment for ESCC.
  13. Receipt of a live vaccine within 28 days prior to first study drug administration.

      NOTE: Seasonal vaccines for influenza are generally inactivated vaccines and are allowed. Intranasal vaccines are live viruses and are not allowed.
  14. Has any of the following cardiovascular risk factors:

      * Ongoing cardiac chest pain, defined as moderate pain that limits instrumental activities of daily living.
      * Symptomatic pulmonary embolism within 28 days of the first study drug administration.
      * Any history of acute myocardial infarction within 6 months of the first study drug administration.
      * Any history of heart failure meeting New York Heart Association (NYHA) Classification III or IV within 6 months before first study drug administration.
      * Any event of ventricular arrhythmia > Grade 2 in severity within 6 months before first study drug administration.
      * Any history of cerebrovascular accident or transient ischemic attack within 6 months before first study drug administration.
      * Uncontrolled hypertension: systolic pressure ≥ 160 mmHg or diastolic pressure ≥ 100 mmHg despite anti-hypertension medications ≤ 28 days before randomization or first dose of study drug.
      * Left ventricular ejection fraction (LEVF) < 50%.
      * QTc interval calculated according to the Fridericia standard, > 450 msec for male and > 470 msec for female.
      * Any episode of syncope or seizure ≤ 28 days before first study drug administration.
  15. Patients with other poorly controlled concomitant diseases, such as chronic obstructive pulmonary disease (COPD), asthma, interstitial lung disease.
  16. Patients with a history of HIV (HIV antibody positive), or uncontrolled infection with hepatitis B or hepatitis C infection, or diagnosis of immunodeficiency that is related to, or results in chronic infection.

      * Patients with known hepatitis B virus (HBV) who have controlled infection (serum hepatitis B virus DNA polymerase chain reaction (PCR) that is below the limit of detection AND receiving anti-viral therapy for hepatitis B) are permitted.
      * Patients with hepatitis C virus (HCV) antibody positive but have controlled infection (undetectable HCV RNA by PCR either spontaneously or in response to a successful prior course of anti-HCV therapy) are permitted.
  17. BMI≤18.5 kg/m2.
  18. Known active alcohol or drug abuse or dependence.
  19. Any other circumstances that the investigator considered inappropriate for participation in the study, or that would interfere with the assessment of safety and effectiveness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-06-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | From the signing of the ICF through 90 days after the last dose
  Incidence and severity of adverse events (AEs), immune-related adverse events (irAEs), serious adverse events (SAEs) assessed by NCI-CTCAE v5.0, based on testing results of vital signs, physical examinations, 12-lead ECG and laboratory tests as well as participants reported adverse events.
PK parameter | 1 hour prior to the first and the sixth dose of IPM514, and 2h(±5min）、6h (±5min), 24h (±30min), 48h(±2h) hours post the first and the sixth dose of IPM514.
  The time to peak (Tmax) will be analyzed by quantitative PCR (qPCR) for mRNA in peripheral blood
PK parameter | 1 hour prior to the first and the sixth dose of IPM514, and 2h(±5min）、6h (±5min), 24h (±30min), 48h(±2h) hours post the first and the sixth dose of IPM514.]
  The maximum concentration (Cmax) will be analyzed by quantitative PCR (qPCR） for mRNA in peripheral blood
PK parameter | 1 hour prior to the first and the sixth dose of IPM514, and 2h(±5min）、6h (±5min), 24h (±30min), 48h(±2h) hours post the first and the sixth dose of IPM514.
  The half-life (T1/2) will be analyzed by quantitative PCR (qPCR) for mRNA in peripheral blood
PK parameter | 1 hour prior to the first and the sixth dose of IPM514, and 2h(±5min）、6h (±5min), 24h (±30min), 48h(±2h) hours post the first and the sixth dose of IPM514.
  The area under the curve (AUC) will be analyzed by quantitative PCR (qPCR) for mRNA in peripheral blood

SECONDARY OUTCOMES:
ORR | up to 49 weeks
  The ORR was defined as the percentage of participants in the study whose best overall response was either CR or PR as assessed by investigators based on RECIST v 1.1 and iRECIST.
PFS | up to 49 weeks
  PFS was defined as the time from the date of first study dose to disease progression or death whichever occurs first.
DCR | up to 49 weeks
  The DCR was defined as the percentage of participants who achieve CR, PR, and SD based on RECIST v 1.1 and iRECIST.
DOR | up to 49 weeks
  DOR for responders (CR or PR) was defined as the time interval between the date of the earliest qualifying response and the date of progressive disease or death for any cause, whichever occurred earlier.
Number Of Participants With Anti-drug Antibodies (ADAs) | within 1 hour prior to the 1st, 6th and 8th administration of IPM514
  The immunogenicity will be evaluated via the incidence and titer of anti-drug antibodies (ADAs)